

#### Statistical Analysis Plan

NCT Number: NCT05382104

Title: A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food on Maribavir (TAK-620) Pharmacokinetics in Healthy Adult Participants

Study Number: TAK-620-1025

Document Version and Date: Original Version (15-June-2022)

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.



#### STATISTICAL ANALYSIS PLAN

Study Number: TAK-620-1025

Phase: 1
Version: Final
Date: 15-June-2022

Biometrics

Plant Phase: 1

Plant Phase: 1

Version: Final
Date: 15-June-2022 A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food on Maribavir (TAK-620) Pharmacokinetics in Healthy Adult Participants

Prepared by:

Data Management and Biometrics

Celerion

MS

Clinical Pharmacology and Pharmacometrics

**Data Management and Biometrics** 

Celerion

Based on:

Protocol Version: Original

Protocol Date: 27-Apr-2022

#### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.

 15-June-2022

#### **REVISION HISTORY**

| Version | Approval Date | Primary Rationale for Revision |
|------------------|---------------|--------------------------------|
| Original Version | 15-June-2022 | Not Applicable |

For non-commercial use only

#### **Approval Signatures**

Electronic signature can be found on the last page of this document.

Study Title: A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the

Effect of Food on Maribavir (TAK-620) Pharmacokinetics in Healthy

**Adult Participants** 



#### **TABLE OF CONTENTS**

| 1.0 | ( | OBJEC | TIVES, ENDPOINTS AND ESTIMANDS | 8 |
|-----|-----|-------|---------------------------------------------------|----|
| | 1.1 | Obj | ectives | 8 |
| | | 1.1.1 | Primary Objectives | 8 |
| | : | 1.1.2 | Secondary Objective | 8 |
| | | 1.1.3 | Exploratory Objective | 8 |
| | 1.2 | Enc | lpoints | 8 |
| | | 1.2.1 | Primary Endpoints | 8 |
| | : | 1.2.2 | Secondary Endpoints | 8 |
| | | 1.2.3 | Exploratory Endpoints | 9 |
| | 1.3 | Esti | imand(s) | 9 |
| 2.0 | | STUDY | Y DESIGN | 10 |
| 3.0 | , | STATI | STICAL HYPOTHESES AND DECISION RULES | 11 |
| | 3.1 | Stat | tistical Hypotheses | 11 |
| | 3.2 | Stat | tistical Decision Rules | 11 |
| | 3.3 | Mu | ltiplicity Adjustment | 11 |
| 4.0 | , | SAMPl | LE-SIZE DETERMINATION | 11 |
| 5.0 | 1 | ANAL | YSIS SETS | 12 |
| | 5.1 | PK | tistical Hypotheses | 12 |
| | 5.2 | Saf | ety Set | 12 |
| 6.0 | | STATI | STICAL ANALYSIS | 12 |
| | 6.1 | Ger | neral Considerations | 12 |
| | ( | 6.1.1 | Handling of Treatment Misallocations | 14 |
| | 6.2 | Stu | dy Information | 14 |
| | 6.3 | Dis | position of Participants | 14 |
| | 6.4 | Der | mographic and Other Baseline Characteristics | 14 |
| | ( | 6.4.1 | Demographics | 14 |
| | ( | 6.4.2 | Medical History and Concurrent Medical Conditions | 14 |
| | 6.5 | Me | dication History and Concomitant Medications | 15 |
| | 6.6 | Eff | icacy Analysis | 15 |
| | 6.7 | Saf | ety Analysis | 15 |
| | ( | 6.7.1 | Adverse Events | 15 |
| | ( | 6.7.2 | Adverse Events of Special Interest | 16 |
| | ( | 6.7.3 | Clinical Laboratory Evaluation | 16 |
| | ( | 6.7.4 | Vital Signs | 18 |

| TAK-620-1<br>Statistical A | 025<br>Analysis Plan | <br>15-June-2022 |
|---|---|---|
| 6.7 | 7.5 12-Lead ECG | 19 |
| 6.7 | 7.6 Physical Examinations | 19 |
| 6.7 | 7.7 Overdose | 19 |
| 6.7 | 7.8 Extent of Exposure and Compliance | |
| 6.8 | Pharmacokinetic Analyses | |
| 6.8 | 8.1 Food-effect Estimation | 20 |
| 6.8 | 8.2 Non-Parametric Analysis | 21 |
| 6.8 | 8.3 Exploratory Analysis | |
| 6.9 | Patient Reported Outcomes (PROs) and Health Care Utilization | |
| | Analysis | |
| 6.10 | Preliminary Analyses | 21 |
| 6.11 | Interim Analyses | 21 |
| 6.12 | Data Monitoring Committee/Internal Review Committee/ [Oth | |
| 7.0 RF | Committees] | 22 |
| 8.0 CH | HANGES TO PROTOCOL PLANNED ANALYSES | 22 |
| 9.0 AI | PPENDIX | 23 |
| 9.1 | Changes From the Previous Version of the SAP | 23 |
| 9.2 | Data Handling Conventions | 23 |
| 9.3 | Data Handling Conventions | 25 |
| LIST OF | IN-TEXT TABLES Study Schematic | |
| Table 2.a | Study Schematic | 10 |
| Table 2.b | Study Treatments for Study Investigational Drug | |

TAK-620-1025  Statistical Analysis Plan 15-June-2022

#### ABBREVIATIONS

AE adverse event

AUC<sub>12</sub> area under the concentration-time curve, from time 0 to 12

 $AUC_{\infty}$  area under the concentration-time curve, from time 0 to infinity, calculated using the

observed value of the last quantifiable concentration

AUC<sub>extrap%</sub> area under the curve from the last quantifiable concentration to infinity calculated using the

observed value of the last quantifiable concentration, expressed as a percentage of AUC∞

AUC<sub>last</sub> area under the concentration-time curve, from time 0 to the time of the last quantifiable

concentration

BLQ below the limit of quantitation

BMI body mass index

C<sub>12</sub> concentration at 12 hours postdose

CI confidence interval

CL/F apparent clearance after oral administration, calculated using the observed value of the last

quantifiable concentration

percent coefficient of variation

C<sub>max</sub> maximum observed concentration

COVID-19 Coronavirus disease 2019

CPAP clinical pharmacology analysis plan

CRF case report form
CRU clinical research unit
CS clinically significant
CSR clinical study report
CV coefficient of variation

DMP data management plan ECG electrocardiogram ET early termination

CV%

Geom CV% geometric coefficient of variation

Geom Mean geometric mean
GI gastrointestinal

GMR geometric mean ratio
ICF informed Consent Form
ID investigational drug
LLN lower limit of normal
LSM least-squares mean
Mean arithmetic mean

MedDRA® Medical Dictionary for Regulatory Activities®

n number of observations

NCA non-compartmental analysis

PCS potentially clinically significant

PK pharmacokinetic(s)

TAK-620-1025  Statistical Analysis Plan 15-June-2022

PT preferred term

QTcF QT interval corrected for heart rate using Fridericia's formula

SAE serious adverse event SAP statistical analysis plan SD standard deviation

**SEM** standard error of the mean

SOC system organ class

terminal disposition phase half-life  $t_{1/_{2}Z}$ **TEAE** treatment-emergent adverse event

TFL tables, figures and listings

lag time to first quantifiable concentration in plasma  $t_{lag}$ 

time to first occurrence of C<sub>max</sub>  $t_{max}$ 

ULN upper limit of normal

apparent volume of distribution during the terminal disposition phase after oral  $V_z/F$ ralue (

administration, calculated using the observed value of the last quantifiable concentration

WHO World Health Organization

 $\lambda_z$ terminal disposition phase rate constant

#### 1.0 OBJECTIVES, ENDPOINTS AND ESTIMANDS

#### 1.1 Objectives

#### 1.1.1 Primary Objectives

To assess the relative bioavailability of a single oral dose of 400 mg maribavir commercial (marketed) tablet formulation administered with a low-fat/low-calorie meal relative to administration under fasting conditions.

To assess the relative bioavailability of a single oral dose of 400 mg maribavir commercial (marketed) tablet formulation administered with a high-fat/high calorie meal relative to administration under fasting conditions.

#### 1.1.2 Secondary Objective

To evaluate the safety and tolerability of a single oral dose of 400 mg maribavir commercial (marketed) tablet formulation when administered under fasting conditions, with a low-fat/low-calorie meal and with a high-fat/high-calorie meal.

#### 1.1.3 Exploratory Objective

To evaluate other pharmacokinetic (PK) parameters of a single oral dose of 400 mg maribavir commercial (marketed) tablet formulation when administered under fasting conditions, with a low-fat/low-calorie meal and with a high-fat/high-calorie meal.

#### 1.2 Endpoints

#### 1.2.1 Primary Endpoints

The following PK parameters in plasma will be analyzed for maribavir:

- *Maximum observed concentration (C<sub>max</sub>)*
- Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC<sub>last</sub>)
- Area under the concentration-time curve from time 0 to infinity, calculated using the observed value of the last quantifiable concentration ( $AUC_{\infty}$ )

#### 1.2.2 Secondary Endpoints

- Treatment-emergent adverse events (TEAEs) and their number, severity, seriousness, and causality
- Changes in vital signs, electrocardiograms (ECGs), and clinical laboratory results (hematology, chemistry, and urinalysis) from baseline to post-baseline time points, and evaluation of clinical signs.

#### 1.2.3 Exploratory Endpoints

Exploratory PK endpoints include (if applicable, but are not limited to) additional PK parameters for maribavir as follows:

- Concentration at 12 hours postdose  $(C_{12})$
- Area under the concentration-time curve from time 0 to 12 ( $AUC_{12}$ )
- Time to first occurrence of  $C_{max}$  ( $t_{max}$ )
- Area under the curve from the last quantifiable concentration to infinity, calculated using the observed value of the last quantifiable concentration, expressed as a percentage of AUC<sub>∞</sub> (AUC<sub>extrap%</sub>)
- Terminal disposition phase rate constant  $(\lambda_z)$
- *Terminal disposition phase half-life*  $(t_{1/2})$
- Apparent volume of distribution during the terminal disposition phase after oral administration, calculated using the observed value of the last quantifiable concentration (V<sub>z</sub>/F)
- Apparent clearance after oral administration, calculated using the observed value of the last quantifiable concentration (CL/F)
- Lag time to first quantifiable concentration in plasma  $(t_{lag})$

#### 1.3 Estimand(s)

Not applicable

#### 2.0 STUDY DESIGN

This is a single-center, open-label, single-dose, randomized, 3-period, 6-sequence, crossover study in healthy adult participants.

Study schematic and dose regimens are shown in Table 2.a and Table 2.b.

**Table 2.a** Study Schematic

| Pretreatment | Predose<br>Assessments | Treatment Per | riods 1-2-3 (a) | Study Exit | Follow-up (b) |
|---|---|---|---|---|---|
| Screening | Check-in | Dosing and Safety and PK Assessments | Safety and PK<br>Assessments | Day 2 of | 7 (±4) days |
| Day -28 to<br>first dosing of<br>ID | Day -1 of<br>Treatment<br>Period 1 | Day 1 | Day 2 | Treatment Period 3 | after last dose |
| | | <b>←</b> Confinement (c) | | | |

<sup>(</sup>a) There will be a washout period of a minimum of 72 hours between each investigational drug (ID) dosing.

Table 2.b Study Treatments for Study Investigational Drug

| | <u> </u> | , , | | |
|---|---|---|---|---|
| Treatment | Investigational Drug | Dose | Dose Regimen | Days on<br>Investigational Drug |
| Treatment A | Maribavir commercial (marketed) tablet formulation | 400 mg (2 x 200-mg) | Single dose, oral, fast | Day 1 |
| Treatment B | Maribavir commercial (marketed) tablet formulation | 400 mg (2 x 200-mg) | Single dose, oral, fed:<br>following a low-<br>fat/low-calorie meal | Day 1 |
| Treatment C | Maribavir commercial<br>(marketed) tablet<br>formulation | 400 mg (2 x 200-mg) | Single dose, oral, fed:<br>following a<br>high-fat/high-calorie<br>meal | Day 1 |

A single dose of 400 mg maribavir (commercial [marketed] tablet formulation) will be administered orally under 3 different feeding conditions:

- 1) Fasting (Treatment A),
- 2) Fed following a low-fat/low-calorie meal (Treatment B), and

<sup>(</sup>b) The clinical research unit (CRU) will contact all participants (including participants who terminate the study early) 7  $(\pm 4)$  days after the last ID administration by telephone or other methods per CRU standards to determine if any AE has occurred or concomitant medications have been taken since the last study visit. If clinically significant findings are observed upon discharge, participants may return to the CRU for re-evaluation per Investigator's discretion.

<sup>(</sup>c) Participants will start the confinement on Day -1 of Treatment Period 1 and will remain confined until Day 2 of Treatment Period 3. Participants may be admitted earlier for Coronavirus disease 2019 (COVID-19) testing not related to study protocol as per CRU requirements.

*3)* Fed following a high-fat/high-calorie meal (Treatment C).

There will be a washout period of a minimum of 72 hours between each ID dosing.

PK samples will be collected predose and up to 36 hours postdose in each treatment period.

Safety and tolerability will be assessed throughout the study by TEAEs, vital signs, ECGs, and clinical laboratory evaluations.

The CRU will contact all participants (including participants who terminate the study early) 7 ( $\pm$  4) days after the last ID administration by telephone or other methods per CRU standards to determine if any AE has occurred or concomitant medications have been taken since the last study visit. If clinically significant findings are observed upon discharge, participants may return to the CRU for re-evaluation per Investigator's discretion.

# .OL only STATISTICAL HYPOTHESES AND DECISION RULES 3.0

#### 3.1 **Statistical Hypotheses**

Not applicable.

#### 3.2 **Statistical Decision Rules**

Not applicable.

#### **Multiplicity Adjustment** 3.3

Not applicable.

#### SAMPLE-SIZE DETERMINATION 4.0

A total of 24 participants should complete all treatment periods of the study.

Sample size calculations were performed using R package PowerTOST and were based on the *following:* 

- The intra-participant coefficient of variation (CV) was assumed at 0.166 and 0.218, respectively for  $AUC_{\infty}$  and  $C_{max}$ , which were estimated from the 90% confidence intervals (CIs) of the geometric mean ratio (GMR) of  $AUC_{\infty}$ , and  $C_{max}$  in Study 1263-104.
- Reference data set is  $AUC_{\infty}$  or  $C_{max}$  under fasting conditions; test data set is  $AUC_{\infty}$  or  $C_{max}$  under fed conditions
- Assumed GMR for Test / Reference: 0.80, 0.85, 0.90, 0.95, or 1.00
- The estimated 90% CI of the GMR at 0.90, with N = 24, is within (0.80, 1.25) for both  $AUC_{\infty}$  and  $C_{max}$

Accounting for possible dropouts, a total of 30 participants will be enrolled.

#### 5.0 ANALYSIS SETS

#### **5.1 PK Set**

All participants who received at least 1 dose of maribavir, did not vomit or had diarrhea within 4 hours of the ID dosing, and have 5 or more postdose time points with evaluable postdose maribavir concentration values that enable non-compartmental analysis (NCA).

Details on criteria for excluding participants from the PK analysis will be described in the Clinical Pharmacology Analysis Plan (CPAP).

#### 5.2 Safety Set

All participants who receive at least 1 dose of maribavir will be included in the safety evaluations.

#### 6.0 STATISTICAL ANALYSIS

#### 6.1 General Considerations

All PK analyses will be conducted using Phoenix<sup>®</sup> WinNonlin<sup>®</sup> Version 8.3.4, or higher. All statistical analyses will be conducted using SAS<sup>®</sup> Version 9.4 or higher. All data recorded on the case report form (CRF) will be listed by participant. All tables, figures, and listings (TFL) shells and numbering list will be included and specified in the TFL shells document.

All concentration and PK parameter data and their descriptive statistics (with the exception of the number of observations) will be presented to 3 significant digits. The number of observations (n) will be presented as an integer (no decimal places).

Concentration values below the lower limit of quantitation (BLQ) will be presented as 'BLQ' in the concentration table listings and footnoted accordingly. BLQ values will be treated as zero for the calculation of summary statistics, the generation of concentration plots, and in the calculation of PK parameters, unless they are deemed questionable (e.g., BLQ value between measurable values), in which case they will be treated as missing and excluded from the concentration summary statistics and the PK analysis. Missing concentration data will not be imputed.

A participant's PK parameter data will be included in the listings but may be excluded from the descriptive summary and statistical model if one or more of the following criteria are met:

- A predose (0 hr) concentration is greater than 5% of that participant's maximum concentration value in that period
- A participant did not meet inclusion/exclusion criteria that may have an effect on the PK
  (as determined by the Takeda Clinical Pharmacology Lead and Celerion Pharmacokinetic
  Scientist)
- A participant vomits or has diarrhea within 4 hours of dosing
- A participant that has less than 5 postdose timepoint with evaluable postdose maribavir concentration values

 A participant deviates substantially from the protocol defined study procedures including but not limited to dosing, dose timing, sample collection, meal timing, etc. (as determined by the Takeda Clinical Pharmacology Lead and Celerion Pharmacokinetic Scientist)
 Note: additional details for excluding participants and/or PK parameters will be detailed in the CPAP.

The details on PK parameter calculations (individual PK parameters for each participant for each period) and TFLs will be outlined in the CPAP and TFL Shells document, as applicable, including specifics on the following:

- Insufficient data to determine a reliable  $t_{1/2z}$  value and other  $\lambda_z$ -dependent parameters
- PK parameters presented by treatment, including the units, precision, and summary statistics that will be presented in in-text and end-of-text tables
- Concentration data presented by treatment, including the units, precision, and summary statistics that will be presented in end-of-text tables
- Concentration data file used for PK analysis
- PK parameter WinNonlin® output file used to generate the TFLs
- PK parameter ratios for  $C_{max}$ ,  $AUC_{last}$ , and  $AUC_{\infty}$ , for each comparison of interest presented in end-of-text tables
- Linear mixed-effects model results presented in in-text and end-of-text tables
- Nonparametric analysis of t<sub>max</sub> and t<sub>lag</sub> for each comparison of interest presented in endof-text tables
- Arithmetic mean concentration-time figures presented as in-text and end-of-text figures
- Individual concentration-time figures and listings presented in Appendices 16.2.6 and 16.2.5, respectively of the clinical study report (CSR)

Safety data will be summarized by randomized treatment sequence or by treatment and time point, as applicable. For the categorical variables, the count and percentages of each possible value will be tabulated, where applicable. The denominator for the percent calculation will be the number of non-missing observations in the safety set for each treatment or sequence. Counts and percentages will be presented as integers. For continuous variables, n, mean, SD, minimum, median, and maximum values will be tabulated. The level of precision will be presented as follows: minimum/maximum in the same precision as in the database, mean/median in one more precision level than minimum/maximum, SD in one more precision level than mean/median, and n will be presented as an integer.

Baseline, unless specified otherwise, is defined as the last observation prior to dosing in each period.

#### **6.1.1** Handling of Treatment Misallocations

Participants with misallocated treatments will be analyzed per the treatment they received rather than per the treatment regimen to which they were randomized.

#### **6.2** Study Information

An overall study information table will be generated including the following items: date of first participant's signed informed consent form (ICF), date of first dose of ID, date of last dose of ID, date of last participant's last visit/contact, date of last participant's last procedure for collection of data for primary endpoint, the version of Medical Dictionary for Regulatory Activities (MedDRA®), the version of World Health Organization (WHO) Dictionary, and SAS version used for creating the datasets.

#### 6.3 Disposition of Participants

Disposition of participants (number of participants dosed, completed the study, discontinued from the study and/or ID, and reason(s) for discontinuation(s)) will be summarized by randomized treatment sequence and overall. Study completion status, including reason for discontinuation of ID and/or study, will be listed by participant.

#### 6.4 Demographic and Other Baseline Characteristics

#### 6.4.1 Demographics

Demographic and baseline characteristics will be summarized by randomized treatment sequence and overall based on the safety set. Summary statistics (n, mean, SD, minimum, median, and maximum) will be generated for continuous variables (age, weight, height, and body mass index [BMI]) and the number and percentages of participants within each category will be presented for categorical variables (sex, race, and ethnicity). Height, weight, and BMI measured at screening will be used in the summaries. Demographic data will also be listed as recorded on the CRF, including the date of informed consent and protocol version.

#### 6.4.2 Medical History and Concurrent Medical Conditions

Medical history to be recorded will include determining whether the participant has any significant conditions or diseases that resolved at or before signing the ICF. All medical history reported by the participant will be recorded regardless of when it may have occurred. Concurrent medical conditions are those significant ongoing conditions or diseases that are present at signing the ICF. Each participant's medical history and concurrent medical conditions will be listed.

Any medical condition starting or worsening after taking the first dose of ID will be classified as a TEAE. All medical history will be coded using MedDRA® version specified in the data management plan (DMP). If available, the medical history and concurrent medical condition listings will include the coded term (preferred term and system organ class [SOC]), start date (if known) and end date (if known) or whether the condition was ongoing, and a description of the condition or event. No summaries or statistical analysis will be performed for these data.

#### 6.5 Medication History and Concomitant Medications

Medication history to be obtained includes any relevant medication stopped at or within 28 days prior to signing the ICF. Concomitant medication includes any medication other than ID taken at any time between first dosing and the end of the study (including follow-up contact). All medication history and concomitant medications recorded during the study will be coded with the WHO Drug Dictionary version specified in the DMP and listed. If available, the listings will include the medication name, coded term, dosage, route of administration, start date and time (if known), end date and time (if known), or whether it continued after study completion, and indication for use. No summaries or statistical analysis will be performed for these data.

#### 6.6 Efficacy Analysis

Not applicable.

#### 6.7 Safety Analysis

Safety will be evaluated by the incidence of TEAEs, severity and relationship(s) of TEAEs, and changes from baseline in the participants' clinical laboratory results, vital signs, and 12-lead ECGs using the safety set. Potentially clinically significant (PCS) laboratory, vital signs, and ECG results will be tabulated. Clinically significant laboratory values, vital signs, and ECGs will be reported as AEs, as applicable. All safety data will be listed by participant, treatment, and assessment time points, including rechecks, unscheduled assessments, and early termination (ET), chronologically.

Continuous variables will be summarized using n, mean, SD, minimum, median, and maximum. Frequency counts and percentages will be reported for categorical data when appropriate. Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators. Postdose recheck, unscheduled, or early termination results will not be used in summaries.

Tables summarizing safety data by assessment time point will only include summaries for baseline and post-baseline time points.

#### **6.7.1** Adverse Events

All AEs captured in the database will be listed in by-participant data listings including verbatim term, coded term, severity (mild, moderate, severe), relationship to ID (related or not related), relationship to COVID-19 and COVID-19 vaccine, frequency, and action relative to the ID as recorded in the CRF. Study procedure taken due to AE will also be listed. All AEs occurring during this study will be coded using the MedDRA® version specified in the DMP. Only TEAEs will be summarized.

A TEAE is defined as an AE that is starting or worsening at the time of or after the first dose of ID administered in the study. Each TEAE will be attributed to the treatment prior to and the closest to the AE based on the AE onset date and time.

If the onset time of an AE is missing and the onset date is the same as a treatment dosing date, then the AE will be counted under the treatment given on the same day. If onset time of an AE is missing and the onset date does not fall on a dosing date, then the AE will be considered treatment emergent for the most recent treatment administered. If the onset date of an AE is missing, then the AE will be considered treatment emergent and attributed to the first treatment received. If severity is missing, the AE will be counted as severe, and if relationship is missing, the AE will be counted as related.

TEAEs will be tabulated by treatment (including overall), SOC, and preferred term. Summary tables will include number of participants reporting the TEAE as percent of safety set by treatment and overall. The most commonly reported non-serious TEAEs (i.e., those events reported by >5% of participants in any treatment, excluding serious adverse events (SAEs) will also be summarized. The denominators for percent calculations will be the number of participants dosed for each treatment. In addition, TEAEs will be summarized as number of TEAEs and percentage of TEAEs for each treatment and overall.

Additional TEAE summary tables will be presented by severity and relationship to ID. If a participant has multiple TEAEs with different severity levels within the same preferred term (PT), the participant will be counted in the most severe category only. For relationship to ID, if a participant has both related and unrelated TEAEs with the same PT, the participant will be counted as having related TEAEs.

An overview summary of TEAEs table, including number of participants with TEAEs, SAEs, treatment-related TEAEs, treatment-related SAEs, TEAEs by severity, and AEs leading to discontinuation will be provided.

Should any SAEs (including all-cause mortalities) occur, they will be summarized the same way as TEAEs. All AEs will be displayed in the data listings and TEAEs will be discussed in the text of the CSR.

#### 6.7.2 Adverse Events of Special Interest

Adverse events of special interest will be identified in the data listings, and will be discussed in the CSR, but will not be summarized separately. Adverse events of special interest for maribavir include dysgeusia and gastrointestinal (GI)-related events.

#### 6.7.3 Clinical Laboratory Evaluation

Clinical laboratory tests will be measured as described in Table 6.a:

Table 6.a Collection of Laboratory Samples

| Clinical Laboratory<br>Panels | Time Point | | |
|---|---|---|---|
| | Period | CRF/Listing Day and Hour | Table |
| | Screening | | NA |

TAK-620-1025 Statistical Analysis Plan

 15-June-2022

| Clinical Laboratory Panels | Time Point | | |
|---|---|---|---|
| | Period | CRF/Listing Day and Hour | Table |
| | 1 | Day -1 PRE-DOSE | Baseline |
| Serum Chemistry,<br>Hematology, Urinalysis | 2 | Day 1 PRE-DOSE | Period 2 Predose |
| | 3 | Day 1 PRE-DOSE<br>Day 2 Hour 24 | Period 3 Predose<br>Period 3 Day 2 |

Time points in the CRF/Listing column are approximated/based on the blank CRF and it should be noted that the data listings will reflect the data found in the final participant CRFs.

If applicable, an early termination assessment will be performed.

NA = Not Applicable

For all numeric values of laboratory test results, summary statistics (n, mean, SD, minimum, median, and maximum) will be presented at each scheduled visit using the units found in the source data. Change from baseline will be summarized in a similar manner. Baseline is defined as the last assessment including rechecks taken prior to the first dose in Period 1. The mean value calculated for each assessment time point will be compared to the reference range and flagged if outside of the reference range (\* if above the reference range and ^ if below the reference range). In the event there is more than one reference range for a laboratory test, the comparison will be made against the lowest of the lower ranges and the highest of the higher ranges. Postdose unscheduled, recheck, or ET assessments will not be used in summaries. All clinical laboratory data will be listed by participant. Urine drug screen will be performed at screening and check-in, and results will be listed by participant.

Out-of-normal range flags will be recorded as high (H) and low (L) for numerical results and did-not-match (\*) for categorical results. For each laboratory test, a shift table will be developed comparing the frequency and percentage of the results at baseline (above normal (H), normal (N), or below normal (L)) with the postdose time points. For urinalysis tests, the categories are normal (N) and abnormal (A). Out-of-range values and corresponding recheck results will be listed.

If a value fails the reference range, it will automatically be compared to a laboratory clinically significant (CS) range. If the value falls within the CS range, it will be noted as "N" for not clinical significant. If the value fails the CS range, it will be flagged with a "Y" which prompts the investigator to determine how the out-of-range value should be followed using 4 Investigator flags: "N", not clinically significant, "R", requesting a recheck, "^", checking at the next scheduled visit, or "Y", clinically significant. Additionally, the investigator will provide a 4th flag when the 3rd flag indicates "R" or "^". This 4th flag is intended to capture final CS (+)/NCS (-) when the 3rd flag does not document significance.

Individual postdose serum chemistry or hematology results that meet Takeda's PCS criteria, including recheck, unscheduled, and ET results, will be listed and tabulated. A participant's value will be considered PCS if it meets one of the criteria described in Appendix A and if it is worse than the participant's baseline value. The number and percentages of participants with at

least one postdose result considered PCS will be provided. A participant mapping table will also be provided to show which participants with worsened postdose values met each category. All clinical laboratory PCS values will also be listed in by-participant data listings.

#### 6.7.4 Vital Signs

Vital signs will be measured as described in Table 6.b:

Table 6.b Collection of Vital Signs

| Parameter | Time Point | | |
|---|---|---|---|
| | Period | CRF/Listing Day and Hour | Table |
| | Screening | | NA |
| Blood Pressure, Heart<br>Rate | 1, 2, 3 | Day 1 PRE-DOSE<br>Day 2 Hour 24 | Baseline<br>Hour 24 |
| | 3 | Day 2 Hour 36 | Hour 36 |
| Respiration, Temperature | Screening | 10 | NA |
| | 3 | Day 2 Hour 36 | NA |

Time points in the CRF/Listing column are approximated based on the blank CRF and it should be noted that the data listing will reflect the data found in the final participant CRFs.

If applicable, an early termination assessment will be performed.

NA = Not applicable

Summary statistics (n, mean, SD, minimum, median, and maximum) will be presented for vital sign results by treatment and time point. Change from baseline will be summarized in a similar manner. Baseline is defined as the last assessment including rechecks taken prior to dosing in each treatment. Postdose unscheduled or recheck assessments will not be used in analysis. Vital sign data will be listed by participant

Individual postdose vital sign results that meet Takeda's PCS criteria, including recheck, unscheduled, and ET results, will be listed and tabulated. A participant's value will be considered PCS if it meets one of the criteria described in Appendix B and if it is worse than the participant's baseline value. The number and percentages of participants with at least one postdose result considered PCS will be provided. A participant mapping table will also be provided to show which participants with worsened postdose values met each category. All clinical laboratory PCS values will also be listed in by-participant data listings.

 15-June-2022

#### 6.7.5 12-Lead ECG

ECGs will be measured as described in Table 6.c:

Table 6.c Collection of ECG Measurements

| Parameter | Time Point | | |
|---|---|---|---|
| | Period | CRF/Listing Day and Hour | Table |
| | Screening | | NA |
| HR, PR, QRS, QT, QTcF, RR | 1, 2, 3 | Day 1 PRE-DOSE<br>Day 2 Hour 24 | Baseline<br>Hour 24 |
| | 3 | Day 1 Hour 3.5<br>Day 2 Hour 36 | Hour 3.5<br>Hour 36 |

Time points in the CRF/Listing column are approximated/based on the blank CRF and it should be noted that the data listing will reflect the data found in the final participant CRFs.

If applicable, an early termination assessment will be performed.

NA = Not applicable

Summary statistics (n, mean, SD, minimum, median, and maximum) will be presented for ECG results by treatment and time point. Change from baseline will be summarized in a similar manner. Baseline is defined as the last assessment including rechecks taken prior to dosing in each treatment. Postdose unscheduled or recheck assessments will not be used in analysis. ECG data will be listed by participant

Individual postdose ECG results that meet Takeda's PCS criteria, including recheck, unscheduled, and ET results, will be listed and tabulated. A participant's value will be considered PCS if it meets one of the criteria described in Appendix C and if it is worse than the participant's baseline value. The number and percentages of participants with at least one postdose result considered PCS will be provided. A participant mapping table will also be provided to show which participants with worsened postdose values met each category. All clinical laboratory PCS values will also be listed in by-participant data listings.

#### 6.7.6 Physical Examinations

Full physical examinations will be performed at screening and at the end of the study. Additional physical examinations may be performed at other times at the discretion of the Investigator. Physical examination findings will be presented in the data listings by participant.

#### 6.7.7 Overdose

All cases of overdose will be presented in a data listing by participant. Any AEs associated with overdose will be documented.

#### 6.7.8 Extent of Exposure and Compliance

The dates, times, and doses of maribavir will be listed by participant and study period.

CONFIDENTIAL

#### 6.8 Pharmacokinetic Analyses

Blood samples for assessment of plasma maribavir concentrations will be collected as outlined in Table 6.d:

Table 6.d Collection of Blood Samples for Pharmacokinetic Analysis

| Analytes | Matrix | Periods | Scheduled Time (Hours)# |
|---|---|---|---|
| Maribavir | Plasma | 1, 2, and 3 | Predose (0) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, and 36 hours postdose |

<sup>#</sup>The actual date and time of sample collection will be recorded on the source document in the CRF.

Concentrations of plasma maribavir at each sampling time will be listed and summarized descriptively by treatment using the following descriptive statistics: n, mean, SD, CV%, SEM, minimum, median, and maximum. Excluded concentrations will be presented and footnoted as such in the concentration table listings, and those values will be excluded from the descriptive statistics.

Individual participant concentration-time curves will be plotted by treatment on linear and semilog scales. The arithmetic mean profiles of the concentration-time data will be plotted by treatment on linear (with and without SD) and semi-log scales. For arithmetic mean concentration-time plots, the nominal PK sampling times will be used. For individual participant concentration-time plots, the actual PK sampling times will be used.

The PK parameters will be calculated from plasma maribavir concentration-time profiles using NCA methods where all calculations will be based on actual sampling times after maribavir dosing. The PK parameters will be summarized by treatment for each study part using the following descriptive statistics: n, mean, SD, CV%, SEM, minimum, median, maximum, Geom mean, and Geom CV%. Excluded parameters will be presented and footnoted as such in the PK parameter table listings, and those values will be excluded from descriptive statistics.

#### **6.8.1** Food-effect Estimation

A linear mixed-effects model will be applied to In-transformed  $C_{max}$ ,  $AUC_{last}$ , and  $AUC_{\infty}$  with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs will be constructed for the differences between Treatment B (low-fat/low-calorie meal) versus Treatment A (fasting), and Treatment C (high-fat/high-calorie meal) versus Treatment A (fasting). The point estimates and their associated 90% CIs will be then back transformed to provide point estimates and 90% CIs for the ratios of Treatment B (low-fat/low-calorie meal) versus Treatment A (fasting) and Treatment C (high-fat/high-calorie meal) versus Treatment A (fasting).


15-June-2022

The following SAS® code will be used to perform the analysis:

PROC MIXED DATA=xxx;

CLASS SEQUENCE PERIOD TREAT PARTICIPANT;

MODEL LN PARAM = SEQUENCE PERIOD TREAT / DDFM=KR;

RANDOM PARTICIPANT(SEQUENCE);

ESTIMATE "Treatment B vs Treatment A" TREAT -1 1 0 / CL ALPHA=0.1 E;

ESTIMATE "Treatment C vs Treatment A" TREAT -1 0 1 / CL ALPHA=0.1 E;

LSMEANS TREAT;

RUN;

#### **6.8.2** Non-Parametric Analysis

Analysis of t<sub>max</sub> and t<sub>lag</sub> will be performed by nonparametric Wilcoxon Signed-Rank test. This analysis will be based on the PK set. The difference of medians (treatment effect) and the corresponding 90% CI will be estimated using the Hodges-Lehmann method and Walsh Averages. The t<sub>max</sub> and t<sub>lag</sub> parameters will not be ln-transformed. The comparisons of interest are the same as in the linear mixed-effects model.

### **6.8.3** Exploratory Analysis

In a separate analysis, not conducted by Celerion, both non-compartmental and compartmental PK modeling will be used to simulate and to project the steady-state AUC<sub>12</sub>, C<sub>max</sub> and C<sub>12</sub> after theoretical regimens of multiple twice daily (BID) oral doses of 400 mg maribavir commercial (marketed) formulation under different dosing conditions (Treatment A, B, or C). The results from the exploratory analysis will not be listed in the CSR and will be detailed in a separate report.

Additional exploratory analyses may be conducted and reported separately.

# 6.9 Patient Reported Outcomes (PROs) and Health Care Utilization Endpoints Analysis

Not applicable.

#### 6.10 Preliminary Analyses

Preliminary PK analyses will be completed as described in the CPAP and Section 6.8 of the SAP, with the following changes: 1) QCed data will be used (not QAed); 2) nominal times (not actual sampling times) will be used for the calculation of PK parameters; and 3) tables and figures will be created using Phoenix<sup>®</sup> WinNonlin<sup>®</sup> Version 8.3.4 or higher, except for the tables presenting the linear mixed-effects model data which will be generated using SAS<sup>®</sup> Version 9.4 or higher.

#### **6.11** Interim Analyses

Not applicable.

 15-June-2022

# 6.12 Data Monitoring Committee/Internal Review Committee/ [Other Data Review Committees]

Not applicable.

#### 7.0 REFERENCES

Not applicable.

#### 8.0 CHANGES TO PROTOCOL PLANNED ANALYSES

The analyses described in this SAP do not differ from those specified in the protocol.

For non-commercial use only

#### 9.0 APPENDIX

#### 9.1 Changes From the Previous Version of the SAP

Not applicable.

#### 9.2 Data Handling Conventions

PCS values must be more extreme than those seen at baseline (e.g. if the baseline value is below the low abnormal value, then the postdose PCS value must be lower). Safety laboratory, vital sign, and ECG values will be identified as PCS using the following criteria:

# Appendix A Criteria for Identification of PCS Safety Laboratory Values Hematology—Criteria for PCS Values

| Parameter | Unit | Low Abnorma | High Abnormal |
|---|---|---|---|
| Hemoglobin | Conventional | <0.8 × LLN | >1.2 × ULN |
| Hematocrit | Conventional | <0.8 × LLN | >1.2 × ULN |
| RBC count | Conventional | <0.8 × LLN | >1.2 × ULN |
| WBC count | Conventional | <0.5 x LLN | >1.5 x ULN |
| Platelet Count | Conventional | <75 x 10 <sup>9</sup> /L | $>600 \times 10^9/L$ |

LLN=lower limit of normal, RBC=red blood cell, ULN=upper limit of normal, WBC=white blood cell.

# Serum Chemistry—Criteria for PCS Values

| Parameter | Unit | Low Abnormal | High Abnormal |
|----------------------|--------------|--------------|---------------|
| ALT | Conventional | 6 | >3x ULN |
| AST | Conventional | | >3x ULN |
| GGT | Conventional | | >3x ULN |
| Alkaline phosphatase | Conventional | | >3x ULN |
| Total Bilirubin | Conventional | | >1.5x ULN |
| Albumin | Conventional | <2.5 g/dL | |
| Total protein | Conventional | <0.8x LLN | >1.2x ULN |
| Creatinine | Conventional | | >1.5x ULN |
| Blood urea nitrogen | Conventional | | >40 mg/dL |
| Sodium | Conventional | <130 mEq/L | >150 mEq/L |
| Potassium | Conventional | <3.0 mEq/L | >5.3 mEq/L |
| Glucose | Conventional | <50 mg/dL | >300 mg/dL |
| Chloride | Conventional | <75 mmol/L | >126 mmol/L |
| Calcium | Conventional | <7.7 mg/dL | >11.1 mg/dL |
| Bicarbonate | Conventional | <8.0 mmol/L | |

ALT=alanine aminotransferase, AST=aspartate aminotransferase, GGT=γ-glutamyl transferase, LLN=lower limit of normal, ULN=upper limit of normal.

 15-June-2022

## Appendix B Criteria for PCS Values for Vital Signs

| Parameter | Unit | Lower Criteria | Upper Criteria |
|---|---|---|---|
| Heart Rate | bpm | <40 | >115 |
| Systolic blood pressure | mm Hg | <90 | ≥160 |
| Diastolic blood pressure | mm Hg | <50 | ≥100 |
| Systolic blood pressure change from baseline | mm Hg | | >20, >30 |
| Diastolic blood pressure change from baseline | mm Hg | | >20, >30 |

For non-commercial use only

 15-June-2022

## Appendix C Criteria for PCS Values for Electrocardiograms

| Parameter | Unit | Lower Criteria | Upper Criteria |
|------------|------|----------------|----------------------------------------|
| Heart rate | bpm | <40 | >115 |
| PR | msec | ≤80 | ≥200 |
| QRS | msec | ≤80 | ≥180 |
| QTcF | msec | <300 | >500 |
| | | | Or |
| | | | >450 and ≥30 msec change from baseline |

## 9.3 Analysis Software

SAS® Version 9.4 or higher will be used for all statistical analyses provided in the CSR.

For non-commercial use only

#### **Certificate Of Completion**

Envelope Id: 0831B915C21E40999BA40CCCE0F62BB9

Subject: Please DocuSign: CA36719\_(TAK-620-1025)\_SAP\_Final\_15Jun2022.pdf

Department: GIBU

Document Type: Project Plan

Source Envelope: Document Pages: 25 Certificate Pages: 2

AutoNav: Enabled

Envelopeld Stamping: Enabled

Time Zone: (UTC+09:00) Osaka, Sapporo, Tokyo

Status: Completed

**Envelope Originator:** 

40 Landsdowne Street Cambridge, MA 02139

IP Address:

#### **Record Tracking**

Status: Original

6/16/2022 11:04:27 PM

Holder:

Signatures: 1

Initials: 0

Location: DocuSign

#### Signature

Signature Adoption: Pre-selected Style

Signer Events

**Timestamp** 

Sent: 6/16/2022 11:05:49 PM Viewed: 6/16/2022 11:14:16 PM Signed: 6/16/2022 11:14:43 PM

6/16/2022 11:14:43 PM

Takeda - DocuSign GxP

Security Level: Email, Account Authentication (Required)

Signed by link sent to

Signature ID:

Using IP Address:

Security Checked

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

Electronic Record and Signature Disclosure:

Not Offered via DocuSign

Completed

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete | Hashed/Encrypted<br>Security Checked<br>Security Checked | 6/16/2022 11:05:49 PM<br>6/16/2022 11:14:16 PM<br>6/16/2022 11:14:43 PM |

For non-commercial use only